CLINICAL TRIAL: NCT07299032
Title: A Randomized Controlled Study on the Localization Efficiency of Optical Motion Capture-Assisted Ultrasound Pre-localization in Pediatric Extracorporeal Shock Wave Lithotripsy
Brief Title: Optical Motion Capture-Assisted Ultrasound for Pediatric ESWL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Qibo Hu, Resident Physician, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URO-2025-12
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Urolithiasis; Extracorporeal Shock Wave Lithotripsy; Optical Motion Capture; Ultrasound Localization; Randomized Controlled Trial; Localization Efficiency
MeSH Terms: interventions — Lithotripsy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): ESWL with Optical Motion Capture-Assisted Ultrasound Localization
  Interventions: Device: ESWL with Optical Motion Capture-Assisted Ultrasound Localization
- Control Group (Active Comparator): ESWL with Conventional Ultrasound Localization
  Interventions: Device: ESWL with Conventional Ultrasound Localization

INTERVENTIONS:
Device: ESWL with Optical Motion Capture-Assisted Ultrasound Localization — Step 1: The physician holds the ultrasound probe to freely scan the patient's target area. Ultrasound images are displayed in real-time to identify and lock onto the stone's position.
  Step 2: Activate the optical motion capture system. High-speed cameras capture the spatial trajectory of the ultrasound probe, while synchronized AI algorithms recognize the stone image to digitally generate the stone's 3D spatial coordinates.
  Step 3: The system automatically matches the position of the ultrasound probe with the shock wave source. Using preset algorithms, it drives the robotic arm to fine-tune the posture, completing the focal point alignment between the probe and the wave source. This ensures the stone is precisely located at the central focus of the lithotripsy energy. Once localization is complete, relevant equipment parameters are locked.
  Arms: Experimental Group
Device: ESWL with Conventional Ultrasound Localization — 1. The physician performs a freehand ultrasound scan based on clinical experience to locate the stone and verify its position.
  2. The ultrasound probe is secured to the dedicated ultrasound bracket of the Dornier lithotripter. The physician manually adjusts the bracket angle while simultaneously controlling the lithotripter's X, Y, and Z-axis movements. The ultrasound image is repeatedly aligned until the stone is confirmed to be precisely located at the focal point of the shock wave energy. Upon completion of localization, the equipment parameters are locked.
  Arms: Control Group

SUMMARY:
The incidence of pediatric urinary system stones has shown an upward trend in recent years, and Extracorporeal Shock Wave Lithotripsy (ESWL) has become one of the most important minimally invasive treatments for pediatric upper urinary tract stones. Currently, the widely used clinical ultrasound mechanical coupling localization mode suffers from issues such as limited scanning degrees of freedom and difficulty in intuitively grasping the spatial relationship between the stone and the focal point. These issues lead to prolonged stone pre-localization times, significant reliance on operator experience, and a steep learning curve for young and primary care physicians, thereby restricting the standardization and widespread promotion of pediatric ESWL.

Building upon existing ESWL equipment, this project independently constructs an "Optical Motion Capture-Assisted Ultrasound Pre-localization System." By utilizing multi-camera infrared motion capture to acquire the 3D pose of the ultrasound probe and the shock wave source in real-time and establishing a unified spatial coordinate system, the system achieves automatic conversion and visual display of the stone's position from the ultrasound image to the shock wave focal point coordinates. This guides the operator to quickly complete focal point pre-localization after freely scanning for the stone. Results from preliminary phantom studies and initial clinical pilot experiments indicate that, while maintaining the routine ESWL workflow, this system can significantly shorten the first effective pre-localization time for pediatric stones from approximately 15 minutes to around 5 minutes, without a significant decrease in the stone clearance rate. This suggests the technology possesses good engineering feasibility and clinical application prospects.

This study proposes to conduct a single-center, prospective, single-blind randomized controlled clinical trial. Pediatric patients with upper urinary tract stones eligible for ESWL will be randomly assigned 1:1 to an experimental group and a control group. The experimental group will use the Optical Motion Capture-Assisted Ultrasound Pre-localization System for stone pre-localization, while the control group will use the routine ultrasound mechanical coupling localization method.

The **primary outcome measure** is the time to first effective stone pre-localization. **Secondary outcomes** include the stone clearance rate evaluated by imaging at 4 and 12 weeks post-operation, the total number of shock waves released and total energy, total procedure time, intraoperative and postoperative complication rates, sedation/anesthesia dosage, and family satisfaction. Additionally, the study will systematically evaluate the system's impact on physician learning curves and work intensity by analyzing the localization success rate of operators with different seniority levels, learning curves (the trend of localization time versus the number of cases), and subjective workload scores.

The core scientific question this project aims to answer is: Under the premise of not compromising the therapeutic efficacy and safety of pediatric ESWL, can optical motion capture-assisted ultrasound pre-localization significantly improve stone localization efficiency, reduce operator workload, and shorten the learning curve for young physicians, thereby enhancing the standardization and accessibility of pediatric ESWL? The expected results will provide an evidence-based foundation for optimizing pediatric ESWL localization modes and formulating relevant technical standards and training programs. Furthermore, it will lay the clinical validation groundwork for future intelligent lithotripsy systems integrating functions such as intelligent identification and robotic arm automatic tracking.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 0 to 14 years with a confirmed diagnosis of upper urinary tract stones.
* Diagnosis confirmed by ultrasound or low-dose CT; stone long diameter ≤ 20 mm (for upper ureteral stones, diameter ≤ 15 mm); absence of urinary tract structural malformations.
* Meeting the indications for ESWL with no absolute contraindications, and scheduled to undergo ESWL treatment.
* Guardians provide informed consent and voluntarily sign the written informed consent form; willing and able to cooperate with the 4-week postoperative follow-up and related examinations.
* Preoperative assessment reveals no contraindications to ESWL, such as uncontrolled infection, severe coagulation disorders, or severe impairment of cardiopulmonary, hepatic, or renal function.

Exclusion Criteria:

* Presence of absolute contraindications for ESWL: Uncontrolled severe urinary tract infection or sepsis; severe uncorrected coagulopathy or current use of anticoagulant/antiplatelet medications; severe renal impairment (significantly decreased GFR); active severe cardiopulmonary disease rendering the patient unable to tolerate anesthesia or shock wave therapy; or absence of an anatomically safe shock wave path (e.g., due to severe skeletal deformities).
* Stones suspected to be extremely hard or complex: Refractory stones indicated by excessively high CT Hounsfield Units (HU) or ultrasound Shear Wave Elastography (SWE) values > 13.7 kPa; or cystine stones in children > 2 years of age (associated with significantly low ESWL success rates).
* Anatomical or physiological challenges: Severe obesity that compromises ultrasound localization; or patients with a solitary kidney or poor contralateral renal function accompanied by a large stone burden.
* Prior intervention: History of prior ESWL or other lithotripsy procedures at the target site, which may confound the evaluation of therapeutic efficacy.
* Underlying systemic conditions: Comorbid severe metabolic diseases or hereditary stone diseases (e.g., cystinuria) requiring priority comprehensive management.
* Compliance issues: Guardians unable to cooperate with the complete follow-up process, or patients with a high anticipated risk of being lost to follow-up.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Total Duration of Ultrasound Localization Operation | Timed for the entire duration of a single procedure; calculated immediately upon the conclusion of the operation.
  Defined as the total duration from the initiation of ultrasound localization until the complete conclusion of the target therapeutic procedure (core lithotripsy-related operations) and the withdrawal of instruments. This excludes time for preoperative preparation, anesthesia, and basic postoperative care. It is recorded in real-time using a precise timing tool.

SECONDARY OUTCOMES:
Stone Clearance Rate at 4 Weeks Post-operation | Week 4 after completion of ESWL.
  Defined as the proportion of pediatric patients in each group who achieve clinical success in ESWL for the target stone relative to the total number of study cases in that group at 4 weeks post-operation. The determination is primarily based on ultrasound examination results, combined with a comprehensive assessment of the patient's clinical symptoms.
Localization Accuracy of Optical Motion Capture Assistance | Measured and verified immediately upon completion of the localization for a single procedure.
  Calculated by assessing the accuracy on the x, y, and z axes for both the optical motion capture-assisted ultrasound localization and the conventional Dornier lithotripter ultrasound localization. Specifically, it measures the deviation between the localization result and the actual stone position (a deviation of ≤5mm on each axis is defined as "accurate"). The metric is the proportion of cases deemed accurate out of the total number of cases for the respective localization method. Immediately after ultrasound localization, the deviation is verified using the optical capture coordinate system to assess the degree of matching.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China